CLINICAL TRIAL: NCT01805895
Title: Minocycline in Acute Cerebral Hemorrhage (MACH) Trial
Brief Title: A Pilot Study of Minocycline in Intracerebral Hemorrhage Patients
Acronym: MACH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Jeffrey Switzer, Associate Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00000718
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Results first posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-03

CONDITIONS: Intracerebral Hemorrhage
Keywords: Stroke; Acute Intracerebral Hemorrhage; Intracerebral Hemorrhage; Hemorrhagic stroke; Hemorrhage; Minocycline
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Hemorrhagic Stroke; Hemorrhage; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline (Experimental): This intervention arm will receive a total of 5 doses of Minocycline. Dose 1 of Minocycline will be 400mg IV within 12-hours of onset of symptoms. Dose 2 of Minocycline will be 400mg oral, given daily on days 2-5 . Each dose is 24 hours apart.
  Interventions: Drug: Minocycline
- Control (No Intervention): This arm will not receive any minocycline. This arm will receive standard of care treatment.

INTERVENTIONS:
Drug: Minocycline — This arm will receive a total of 5 doses of minocycline. Dose 1 will be 400mg IV within 12-hours of onset of symptoms. Dose 2 will be 400mg oral, given daily on days 2-5 . Each dose is 24 hours apart.
  Other Names: Dynacin, Minocin
  Arms: Minocycline

SUMMARY:
The MACH Trial is a pilot study of 400mg minocycline over five days in acute intracerebral hemorrhage patients. The study will evaluation the safety and efficacy of minocycline in intracerebral hemorrhage patients.

DETAILED DESCRIPTION:
MACH is a randomized trial of minocycline in intracerebral hemorrhage. 24 total subjects will be randomly assigned to minocycline or control (1:1). The first dose will be given intravenously. Subsequent doses will be given orally every 24 hours for a total of five doses. The study will test to see if the medication is safe in intracerebral hemorrhage. The pharmacokinetics of minocycline in intracerebral hemorrhage will be determined and the impact of minocycline on blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Intracerebral hemorrhage documented by CT scan
* The first dose of the drug can be administered within 12 hours of time last known to be at baseline

Exclusion Criteria:

* Allergy to tetracycline antibiotics
* Pregnancy or suspected pregnancy (pregnancy test will be done on women of child-bearing potential)
* Hepatic and/or renal insufficiency (LFT's >3x upper limit of normal; Creatinine >2mg/dL)
* History of intolerance to minocycline
* National Institutes of Health Stroke Scale score of 4 or less
* Glasgow Coma Scale score of 5 or less
* Surgical evacuation of hematoma planned within 24 hours
* Secondary intracerebral hemorrhage resulting from trauma, arteriovenous malformation, aneurysm, tumor or other causes
* Thrombocytopenia (platelet count <75,000/mm3) or coagulopathy (INR >1.4)
* Previously not independent (prestroke modified Rankin scale score >2)
* Suspected of not being able to comply with the study protocol
* Unlikely to be available for 90 day follow-up
* Pre-existing Do Not Resuscitate (DNR) order or indication that a new DNR order will be implemented within the first 48 hours of hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Switzer, DO, Principal Investigator — Augusta University
Locations (1):
- Georgia Health Sciences University, Augusta, Georgia, United States

REFERENCES:
- [Derived] Fouda AY, Newsome AS, Spellicy S, Waller JL, Zhi W, Hess DC, Ergul A, Edwards DJ, Fagan SC, Switzer JA. Minocycline in Acute Cerebral Hemorrhage: An Early Phase Randomized Trial. Stroke. 2017 Oct;48(10):2885-2887. doi: 10.1161/STROKEAHA.117.018658. Epub 2017 Sep 8. PMID 28887388

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Minocycline | Control
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minocycline | Control | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (14.6) | 61.8 (11.5) | 61.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Modified Rankin Scale
Description: A blinded assessor will perform the modified Rankin Scale (this is the full scale name) after 90 days. This will serve as our efficacy endpoint. The scale measures function. It ranges from 0 to 6 with zero reflecting no disability, 1 to 5 increasing degrees of disability and 6 death. Lower numbers reflect preferred outcome. There are no sub scales.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minocycline | Control
Number analyzed (Participants) | 8 | 8
units on a scale | 3.5 (2.3) | 3.7 (1.4)

2. Secondary Outcome: Safety Assessment
Description: Adverse events will be asses for 90 days. This will serve as our safety endpoint.
Time Frame: 90 days
Measure: Number; unit: adverse events
Arm/Group | Minocycline | Control
Number analyzed (Participants) | 8 | 8
adverse events | 0 | 0

ADVERSE EVENTS:
Arm/Group | Minocycline | Control
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No